CLINICAL TRIAL: NCT01181232
Title: A Randomized, Active Control, Parallel Study to Evaluate the Efficacy and Safety of Zolpidem MR (Stilnox CR) Versus Zolpidem (Stilnox) in Patients With Primary Insomnia
Brief Title: A Study to Compare Efficacy and Safety of Zolpidem Modified Release Formulation Versus Zolpidem in Insomnia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STCR-0901-TW
Record Dates: First submitted 2010-08-04; First posted 2010-08-13 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Initiation and Maintenance Disorders; Primary Insomnia
Keywords: insomnia; zolpidem
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MR low-dose group (Experimental)
  Interventions: Drug: Zolpidem MR
- MR high-dose group (Experimental)
  Interventions: Drug: Zolpidem MR
- IR group (Active Comparator)
  Interventions: Drug: Zolpidem IR

INTERVENTIONS:
Drug: Zolpidem MR — oral
  Other Names: Stilnox CR; Ambient CR
  Arms: MR high-dose group; MR low-dose group
Drug: Zolpidem IR — oral
  Other Names: Stilnox
  Arms: IR group

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of zolpidem MR (modified release) compared to zolpidem IR (immediate release) in patients with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary insomnia based on DSM-IV criteria (307.42)
* Written informed consent has been obtained

Exclusion Criteria:

* Patients with sleep apnea syndrome, narcolepsy, presence or suspicion of periodic leg movement or restless leg syndrome
* Patients with hepatic failure, myasthenia gravis, or hypersensitivity to zolpidem
* Patients who are known to be current drug or alcohol abuser or likely to concomitantly consume alcoholic beverages (more than 3 times/week)
* Patients who have received antihistamines or antipsychotics will not allow to discontinue the previous medication throughout the study
* Patients who are pregnant, lactating or intend to become pregnant during the study period
* Patients who have received antidepressants or anxiolytics will not allow to change the dose or discontinue the previous medication throughout the study
* Any clinically significant condition, which in the opinion of the investigator makes the patients unsuitable for the trial
* Participation in any clinical trial within 1 month prior to randomization

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Rest/activity cycles measured by Actigraphy | For 2 weeks (Day 0, Day 7, Day 14)
Total score of Pittsburgh Sleep Quality Index (PSQI) | For 2 weeks (Day 0, Day 7, Day 14)

SECONDARY OUTCOMES:
Physician's clinical global impression (CGI) | For 2 weeks (Day 0, Day 7, Day 14)
Patient's global impression (PGI) | For 2 weeks (Day 0, Day 7, Day 14)
Sleep latency as derived from sleep diary | For 2 weeks (Day 0, Day 7, Day 14)
Number of awakenings as derived from sleep diary | For 2 weeks (Day 0, Day 7, Day 14)
Total sleep time as derived from sleep diary | For 2 weeks (Day 0, Day 7, Day 14)
Wake time after sleep onset as derived from sleep diary | For 2 weeks (Day 0, Day 7, Day 14)
Day time function as assessed by Epworth Sleepiness Scale (ESS) | For 2 weeks (Day 0, Day 7, Day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (2):
- Taiwan (2):
  - Tainan
  - Taipei